CLINICAL TRIAL: NCT06369389
Title: Evaluation of the Real-life Management of Patients Eligible for CAR-T Cell Therapy for Hematologic Malignancies at Toulouse University Hospital
Brief Title: Real-life Management of Patients Eligible for CAR-T Cell Therapy
Acronym: CARAVAGE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ligue contre le cancer, France (Other); Janssen, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0417
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Hemopathy
Keywords: CAR-T cells; real life; care pathways; quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients eligible for CAR-T treatment: Patients eligible for CAR-T treatment for their hemopathy at TOULOUSE University Hospital under early access or marketing authorization or as part of a clinical trial between 01/01/2019 and 31/12/2028
  Interventions: Other: Patients eligible for CAR-T treatment

INTERVENTIONS:
Other: Patients eligible for CAR-T treatment — Patients eligible for CAR-T treatment for their hemopathy at TOULOUSE University Hospital under early access or marketing authorization or as part of a clinical trial between 01/01/2019 and 31/12/2028

SUMMARY:
Adoptive immunotherapy using CAR-T cells is now one of the Advanced Therapy Medicines routinely used for relapsed or refractory lymphoid hemopathies. In 2023, in France, 5 types of CAR-T cells have marketing authorization for 6 different indications. However, these marketing authorizations are based on clinical trials involving a limited number of selected patients. Real-life data are essential for assessing the post-authorization use of these innovative treatments. The French national DESCAR-T registry, promoted by LYSARC and in which Toulouse University Hospital plays an active role, is an international reference for this real-life evaluation. It does not, however, allow precise evaluation of patient-centered indicators and care pathways.

With the increasing number of indications and candidate patients, Toulouse University Hospital, the only healthcare facility authorized in the Western Occitanie region to administer CAR-T cells, is faced with growing hospital needs and longer treatment times. In 2023, this has necessitated the implementation of new ambulatory and inter-facility care pathways in collaboration with the referral centers of the Onco-Occitanie Ouest regional cancer network. The selection of patients for CAR-T cell treatment is based on objective clinical criteria linked to the pathology (histology, morphological localization, size and kinetics of the tumor mass) and the patient (physiological age, performance index, comorbidities, patient choice). Because of their innovative nature, in a difficult psychological and physical context for the patient (refractory disease), CAR-T cell care pathways also need to be evaluated in terms of their "quality of life" dimension. The impact of non-biological determinants (also described as social and territorial inequalities in health) such as place of residence and distance from healthcare provision, marital, economic and social status, has never been explored on the accessibility and progress of the CAR-T cell treatment pathway.

The creation of a registry of patients eligible for CAR-T cells at Toulouse University Hospital will enable these lines of research to be explored on the scale of a region with a population of 3 million.

DETAILED DESCRIPTION:
Ambispective observational cohort: This observational study is monocentric. For each patient, data will be collected during 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for CAR-T treatment for hemopathy at TOULOUSE University Hospital under early access or marketing authorization or as part of a clinical trial between 01/01/2019 and 31/12/2028
* Patient able to understand the purpose and constraints of the research project
* Patient has read the study information leaflet and does not object to the research.

Exclusion Criteria:

* Patient under guardianship, curatorship or safeguard of justice
* Patient objects to the collection of data concerning him/her

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient major eligible for CAR-T treatment for hemopathy at TOULOUSE University Hospital under early access or marketing authorization or as part of a clinical trial between 01/01/2019 and 31/12/2028
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival of patients with hemopathy eligible for CAR-T cell therapy | 5 years
  Overall survival from CAR-T cell injection to all-cause death

SECONDARY OUTCOMES:
Compare progression-free survival and overall survival of patients according to care pathway and type of hemopathy, and investigate clinical and socioeconomic factors associated with better survival | 5 years
  progression-free survival from CAR-T cell injection to date of progression and overall survival from CAR-T cell injection to all-cause death progression-free survival from CAR-T cell injection to date of progression and overall survival from CAR-T cell injection to all-cause death
Evaluate the time taken to treat patients with CAR-T cells | 5 years
  number of days between the multidisciplinary consultation meeting and the injection of CAR-T cells

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BORIES, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, CHU de Toulouse, France

IPD SHARING:
Plan to Share IPD: No